CLINICAL TRIAL: NCT05790889
Title: A Phase IIb Randomised Controlled Trial of the Safety, Immunogenicity and Efficacy of the Blood-stage Malaria Vaccine Candidates RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in Infants Aged 5-17 Months in Burkina Faso.
Brief Title: A Study to Test Experimental Blood Stage Malaria Vaccine in Burkina Faso.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAC091
Record Dates: First submitted 2023-01-16; First posted 2023-03-30 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Rabies Vaccines; Matrix-M

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Control group) (Placebo Comparator): n= 60. Age= 5-17 months Rabies Vaccine administered on Days 0, 28 and 152.
  Interventions: Biological: Rabies vaccine
- Group 2 (Experimental): n=120 Age= 5-17 months First vaccination of RH5.1 10μg with 50μg Matrix-M will be administered on day 0, followed by a second dose administered on Day 28, followed by a third and final dose at Day 152.
  Interventions: Biological: RH5.1 10μg adjuvated with 50μg Matrix-M
- Group 3 (Control Group) (Placebo Comparator): n= 60. Age= 5-17 months Rabies Vaccine administered on Days 0, 28 and 56.
  Interventions: Biological: Rabies vaccine
- Group 4 (Experimental): n=120 Age= 5-17 months First vaccination of RH5.1 10μg with 50μg Matrix-M will be administered on day 0, followed by a second dose administered on Day 28, followed by a third and final dose at Day 56.
  Interventions: Biological: RH5.1 10μg adjuvated with 50μg Matrix-M
- Group 5 (Experimental): n=120 Age= 5-17 months First vaccination of RH5.2-VLP 5μg with 50μg Matrix-M will be administered on day 0, followed by a second dose administered on Day 28, followed by a third and final dose at Day 56.
  Interventions: Biological: RH5.2 5μg adjuvated with 50μg Matrix-M

INTERVENTIONS:
Biological: Rabies vaccine — Vaccine
  Arms: Group 1 (Control group); Group 3 (Control Group)
Biological: RH5.1 10μg adjuvated with 50μg Matrix-M — Vaccine
  Arms: Group 2; Group 4
Biological: RH5.2 5μg adjuvated with 50μg Matrix-M — Vaccine
  Arms: Group 5

SUMMARY:
This is a Phase IIb randomised controlled trial of the safety, immunogenicity and efficacy of the blood-stage malaria vaccine candidates RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in infants aged 5-17 months in Burkina Faso

DETAILED DESCRIPTION:
During the initial recruitment to Groups 1 and 2, participants will be randomised 1:2 to receive vaccination with the rabies control vaccination or RH5.1/Matrix-M.

During recruitment to Groups 3, 4 and 5, participants will be randomised 1:2:2 to receive vaccination with rabies control vaccination, RH5.1/Matrix-M or RH5.2-VLP/Matrix-M Efficacy of vaccination will be assessed by comparing the incidence of malaria cases in the pooled control groups (Groups 1 and 3) to the incidence of malaria in each investigational vaccine group (Groups 2,4 and 5).

There are three study vaccines: the IMP, 10μg RH5.1 adjuvanted with Matrix-M; 5μg RH5.2-VLP and Rabies Vaccine. Participants will receive the first vaccination of RH5.1 10μg with 50μg Matrix-M (Groups 2 and 4) or RH5.2 5μg with 50μg Matrix-M (Group 5). After approximately 4 weeks, a second dose will be administered, followed by a third and final vaccination approximately 4 weeks later (Groups 3-5) or approximately 4 months later (Groups 1-2). Second and third vaccinations will be administered at the same dose of both vaccine and adjuvant as at the initial vaccination and will be given within the window period of 5 months. Volunteers will be followed for 12 months from final vaccination.

The trial is funded by EDCTP grant number RIA2016V-1649-MMVC and by a Wellcome Trust Translational Award (205981/Z/17/Z)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infant aged 5-17 months at the time of first study vaccination
2. Parent/guardian provides signed/thumb-printed informed consent
3. Infant and parent/guardian resident in the study area villages and anticipated to be available for vaccination and follow-up for 12 months following last dose of vaccination.

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
* Clinically significant skin disorder (psoriasis, contact dermatitis etc.), cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness as judged by the PI or other delegated individual.
* Weight-for-age Z score of less than -3 or other clinical signs of malnutrition.
* History of allergic reaction, significant IgE-mediated event, or anaphylaxis to immunization.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Sickle cell disease.
* Clinically significant laboratory abnormality as judged by the study clinician.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Receipt of any vaccine in the 7 days preceding enrolment, or planned receipt of any other vaccine within 7 days following each study vaccination.
* History of vaccination with another malaria vaccine.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Known maternal HIV infection (no testing will be done by the study team).
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (for corticosteroids, this will mean prednisone, or equivalent, ≥0.5 mg/kg/day; inhaled and topical steroids are allowed).
* Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To assess the protective efficacy against clinical malaria of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area for 6 months after the last vaccination. | From 14 days after the third study vaccination until 6 months after the third study vaccination.
  Time to first episode of clinical malaria (defined as the presence of axillary temperature higher than 37.5 degree celsius and P. Falciparum parasite density >5000 asexual forms/µL)
To assess the safety and reactogenicity of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area. | The month following each vaccination and at 6 and 12 months after administration of the final dose of vaccine.
  Occurrence of solicited systemic reactogenicity signs and symptoms via clinic and home visits

SECONDARY OUTCOMES:
To assess the humoral immunogenicity of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area. | Immunology blood samples will be collected at screening, day of vaccination (V) 1, 14 & 28 days post V2, day of V3, 14 days post V3, 2, 6 and 12 months post V3.
  The following measures will be assessed
  * Serum ELISA response:
    1. Quantitative antigen-specific IgG antibody levels (µg/mL readout) over time - analysis of peak responses and longevity; 2. Antigen-specific antibody subclass/isotype measurement; 3. Antigen-specific antibody avidity measurement; In vitro GIA against 3D7 clone P. falciparum parasites using purified total IgG and a single-cycle pLDH readout assay
  * Purified IgG ELISA versus GIA titration "Quality Analysis"
To assess the protective efficacy against clinical malaria of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area for 3 months after the last vaccination. | From 14 days after the third study vaccination until 3 months after the third study vaccination
  Time to first episode of clinical malaria (defined as the presence of axillary temperature ≥37.5°C and P. falciparum parasite density >5000 asexual forms/µL).
To assess the protective efficacy against clinical malaria of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area | For 12 months after the last vaccination
  Occurrence of solicited local reactogenicity signs and symptoms via clinic and home visits
To assess the protective efficacy against asymptomatic P. falciparum infection of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area, by qPCR. | At 6 and 12 months after administration of the final dose of vaccine.
  Efficacy tested by conducting qPCR analysis
To assess the protective efficacy against asymptomatic P. falciparum infection against gametocytaemia of RH5.1 in Matrix-MTM and RH5.2-VLP in Matrix-MTM in 5-17 months old children living in a malaria-endemic area, by qPCR. | At 6 and 12 months post third study vaccination.
  The proportion of participants in each study arm that show presence of parasite density >5000 asexual forms/µL as measured by quantitative reverse-transcriptase PCR PLUS presence of axillary temperature <37.5°C and absence of history of fever within the last 24 hours. The proportion of participants in each study arm that show presence of parasite density >0 asexual forms/µL as measured by quantitative reverse-transcriptase PCR PLUS presence of axillary temperature <37.5°C and absence of history of fever within the last 24 hours.
To assess the protective efficacy against clinical malaria of RH5.1 in Matrix-M and RH5.2-VLP in Matrix-M in 5-17 months old children living in a malaria-endemic area for 12 months after the last vaccination. | From 14 days after the third study vaccination until 12 months after the third study vaccination
  Time to first episode of clinical malaria (defined as the presence of axillary temperature ≥37.5°C and P. falciparum parasite density >5000 asexual forms/µL).
To assess the protective efficacy against gametocytaemia of RH5.1 in Matrix-M and RH5.2-VLP in Matrix-M in 5-17 months old children living in a malaria-endemic area, by qPCR at 2 and 6 months after administration of the final dose of vaccine | At 2 and 6 months post third study vaccination.
  The proportion of participants in each study arm that show presence of gametocytes >0 gametocytes/μL as measured by quantitative reverse-transcriptase PCR.
Efficacy against incident severe anaemia and blood transfusion requirement | From 14 days after the third study vaccination until 6 months after the third study vaccination.
  The proportion of participants in each study arm with documented Hb <5.0 g/dL identified at clinical presentation in association with P. falciparum asexual parasitaemia > 5000 parasites/µL. The proportion of participants in each study arm with documented Hb <5.0 g/dL identified at clinical presentation and requirement for a blood transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Minassian, Principal Investigator — Honorary Consultant and Chief Investigator - Project clinical trials
Locations (1):
- Institut de Recherche en Sciences de la Santé, Siglé, Boulkiemdé Province, Burkina Faso

REFERENCES:
- [Derived] Natama HM, Salkeld J, Some A, Soremekun S, Diallo S, Traore O, Rouamba T, Ouedraogo F, Ouedraogo E, Dabone KCS, Kone NA, Compaore ZMJ, Kafando M, Bonko MDA, Konate F, Sorgho H, Nielsen CM, Pipini D, Diouf A, King LDW, Shaligram U, Long CA, Cho JS, Lawrie AM, Skinner K, Roberts R, Miura K, Bradley J, Silk SE, Draper SJ, Tinto H, Minassian AM. Safety and efficacy of the blood-stage malaria vaccine RH5.1/Matrix-M in Burkina Faso: interim results of a double-blind, randomised, controlled, phase 2b trial in children. Lancet Infect Dis. 2025 May;25(5):495-506. doi: 10.1016/S1473-3099(24)00752-7. Epub 2024 Dec 10. PMID 39672183